CLINICAL TRIAL: NCT06607770
Title: An Exploratory Study of the Safety and Efficacy of Cryoablation in Combination With Karelizumab and Apatinib for the Treatment of Multiple Primary Lung Cancers Without Known Driver Genes
Brief Title: Safety and Efficacy of Cryoablation With Karelizumab and Apatinib for Multiple Lung Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zhou Chengzhi (Other)
Responsible Party: Sponsor-Investigator, Zhou Chengzhi, chief physician, Guangzhou Institute of Respiratory Disease
Organization: Guangzhou Institute of Respiratory Disease (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CROC-24-08
Record Dates: First submitted 2024-09-11; First posted 2024-09-23 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Patients were started on Carrelizumab in combination with Apatinib 2-3 weeks after cryoablation. Karelizumab 200 mg, q3w, and Apatinib 250 mg, qd. Every 3 weeks is a treatment cycle.
  Interventions: Drug: Karelizumab+Apatinib

INTERVENTIONS:
Drug: Karelizumab+Apatinib — Karelizumab 200mg, q3w, and Apatinib 250mg, qd. every 3 weeks as a treatment cycle.

SUMMARY:
The goal of this clinical trial is to explore the safety and efficacy of cryoablation combined with carlizumab and apatinib in multiple primary lung cancer without known driver genes.Main included population criteria:Clinical and pathological diagnosis of multiple primary lung cancer;Three pulmonary nodules were diagnosed initially or before surgery, without lymph node metastasis;Male or female is 18 years old, and 75 years old;Up to one surgical resection treatment with 2 remaining pulmonary nodules, and postoperative pathology confirmed MIA or AIS and so on.The main questions it aims to answer is safety of cryoablation combined with carilizumab and apatinib in multiple primary lung cancer.Participants will take carplus with apatinib started 2-3 weeks after cryoablation. Carelizumab 200mg, q3w, apatinib 250mg, qd. Every 3 weeks is for one treatment cycle. Until PD, intolerable toxicity, death, patient withdrawal or investigator discretion requires termination.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical and pathological diagnosis of multiple primary lung cancers；
2. There were 3 intrapulmonary nodules ≥ the initial diagnosis or preoperative, and there was no lymph node metastasis；
3. The maximum lesion diameter ≤ 3 cm；
4. At most, patients has undergone surgical resection treatment, and there are ≥ 2 remaining intrapulmonary nodules, and the postoperative pathology confirms that it is MIA or AIS；
5. It is estimated that at least 1 measurable lesion meeting RECIST v1.1 criteria will remain after cryotherapy；
6. Male or female≥ 18 years old and ≤ 75 years old；
7. United States Eastern Cooperative Oncology Group Performance Status (ECOG PS) score of 0 or 1；
8. Expected survival ≥ 12 weeks；
9. Vital organ and bone marrow function meets the following requirements:a.Blood routine: absolute neutrophil count (ANC) ≥1.5× 109/L, platelet (PLT) ≥100× 109/L, hemoglobin (HGB) ≥9 g/dL;b.Liver function: serum total bilirubin (TBIL) ≤1.5 times the upper limit of normal (ULN), alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤2.5 times the ULN, serum albumin (ALB) ≥2.8 g/dL;c.Renal function: serum creatinine (Cr) ≤ 1.5 x ULN, or creatinine clearance ≥ 40 mL/min;
10. Subject with subject sexual partner needs to use one medically approved contraceptive measure (such as intrauterine device, birth control pill or condom, etc.) during study treatment and for 6 months after the end of the study treatment period;
11. Subjects must have signed an IRB/IEC-approved written informed consent form in accordance with competent authority and study site guidelines and be able to comply with protocol-specified visits, treatment protocols, laboratory tests, and related procedures.

Exclusion Criteria:

1. Patients with known EGFR mutations, ALK rearrangements;
2. Conditions that cannot be treated with cryoablation: diffuse lesions in both lungs, extensive pleural metastases with large pleural effusions, tumors adjacent to or encircling large mediastinal vessels, etc;
3. Prior receipt of anti-PD-1, anti-PD-L1, anti-CTLA-4 antibodies, or any other antibody or drug targeting T cell co-stimulation or immune checkpoint pathways;
4. Received the following treatments:a.Received systemic anti-tumor therapy such as chemotherapy, targeted therapy, immunotherapy, etc. within 4 weeks prior to randomization;b.Treatment with any investigational drug within 4 weeks prior to randomization;c.Receipt of high-dose immunosuppressive medications (systemic glucocorticoids greater than 10 mg/day of prednisone or its equivalent) within 4 weeks prior to randomization;d.Major surgery (such as open, thoracotomy, or laparotomy, etc.), or unhealed surgical wounds, ulcers, or fractures within 4 weeks prior to randomization.
5. Known or suspected active autoimmune disease (congenital or acquired);
6. Known allogeneic organ transplantation (other than corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
7. Hypersensitivity to any component of the monoclonal antibody preparation;
8. With interstitial lung disease;
9. With other uncontrolled serious medical conditions;
10. Other acute or chronic illness, psychiatric illness, or abnormal laboratory test values that may result in an increase in the risk associated with study participation or study drug administration, or interfere with the interpretation of study results, and the patient is listed as ineligible for this study in the judgment of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
irAEs rate | 3 years
  Incidence of adverse events occurring during treatment

SECONDARY OUTCOMES:
ORR | 3 years
  Proportion of patients whose tumor volume shrinks to a pre-specified value and who can maintain the minimum timeframe requirement, as the sum of the proportion in complete and partial remission
DCR | 3 years
  Number of cases in remission (PR+CR) and stable lesions (SD) after treatment as a percentage of evaluable cases
DOR | 3 years
  the time between the first time a subject in confirmed complete remission (CR) or confirmed partial remission (PR) reaches confirmed complete remission (CR) or confirmed partial remission (PR) and the time of the first disease progression or death of any cause
PFS | 3 years
  Time from start of patient's treatment to disease progression or death from any cause
OS | 3 years
  Time from patient randomization to patient death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Chengzhi Zhou, doctor, Study Director — The First Affiliated Hospital of Guangzhou Medical University,Guangzhou
Locations (1):
- Chengzhi Zhou, Guangzhou, Guangdong, China